CLINICAL TRIAL: NCT01531634
Title: Promoting Recovery Processes in Women Diagnosed With Borderline Personality Disorder Using a Dynamic Cognitive Intervention
Brief Title: Promoting Recovery Processes in Women With Borderline Personality Disorder Using a Dynamic Cognitive Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0010-12-HYMC
Record Dates: First submitted 2012-02-03; First posted 2012-02-13 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; Women; Dynamic Cognitive Intervention; Recovery; Hope Scale
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dynamic Cognitive Intervention Group (Active Comparator): Twelve Meetings of Dynamic Cognitive Intervention.
  Interventions: Behavioral: Dynamic Cognitive Intervention Group
- No Additional Intervention (No Intervention)

INTERVENTIONS:
Behavioral: Dynamic Cognitive Intervention Group — Twelve meetings of a Dynamic Cognitive Intervention group.
  Other Names: DCI
  Arms: Dynamic Cognitive Intervention Group

SUMMARY:
The field of psychiatric rehabilitation focuses on creating a personal narrative and developing coping strategies and environmental supports. The concept of recovery is person-centered and emphasizes the person's ability to change and to live meaningful life. The strengths approach has a central role in the recovery concept, emphasizing the person's abilities and potential. A preserved cognitive ability can be a significant strength in the recovery process.

Research had shown growing support for the use of cognitive-behavioral approaches as the most effective therapy for people with borderline personality disorder, using structured interventions. A central focus in cognitive therapy is the change of maladaptive schemes. The dynamic-cognitive intervention (DCI) is based on the understanding of structural cognitive modifiability and suggests the use of mediated learning in order to enhance sense of competence and develop better psychological coping skills.

The present study will focus on women diagnosed with borderline personality disorder, with normative cognitive ability seen as a strength as opposed to their emotional ability. This study will examine the effects of a Dynamic Cognitive Intervention on recovery measures and on symptoms severity.

The study will include 30 women aged 18-45 years. Participants will be randomly assigned to an intervention group and a control group. All participants will be assessed before and after intervention using Recovery Assessment Scale, Hope Scale and The Brief Symptom Inventory.

The intervention designed for this study is based on the principles of the Dynamic Cognitive Intervention. The intervention tools that will be used include: a. Instrumental Enrichment tools. b. life events analysis. c. Stories, lyrics and movie clips. d. Worksheets. The intervention encompasses 12 sessions of 1.5 hours, with a routine structure.

The results are expected to contribute to the understanding of the impact of a dynamic cognitive intervention in women diagnosed with borderline personality disorder.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age 18 - 45
* Borderline Personality Disorder, by DSM-V

Exclusion Criteria:

* Current Acute Depressive Episode
* Current Psychotic Episode
* Less Than 12 school years
* Non Compliance with therapy
* Dual diagnosis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)

PRIMARY OUTCOMES:
Change in Recovery Assessment Scale | Change from baseline in Recovery Assessment Scale at 12th meeting (6 up to 12 weeks)
  A baseline Recovery Assessment Scale will be used on the first intervention group meeting. Recovery Assessment Scale will be used again on the last (i.e. 12th) intervention group meeting.

SECONDARY OUTCOMES:
Change in Hope Scale | Change from baseline in Hope Scale at 12th meeting (6 up to 12 weeks)
  A baseline Hope Scale will be used on the first intervention group meeting. Hope Scale will be used again on the last (i.e. 12th) intervention group meeting.
Change in Brief Symptom Inventory | Change from baseline in Brief Symptom Inventory at 12th meeting (6 up to 12 weeks)
  A baseline Brief Symptom Inventory will be used on the first intervention group meeting. Brief Symptom Inventory will be used again on the last (i.e. 12th) intervention group meeting.

CONTACTS AND LOCATIONS:
Overall Officials: Orly Tsabar, B.O.T., Principal Investigator — Tel Aviv University
Locations (1):
- Day Center for Mentally Ill, Netanya, Israel

REFERENCES:
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793